CLINICAL TRIAL: NCT02846662
Title: Randomized Clinical Trial to Evaluate the Effectiveness of an Intervention Using Mobile Technology for the Treatment of Depressive Symptoms in People With Diabetes or Hypertension
Brief Title: Effectiveness of a Mobile Technology Intervention for the Treatment of Depression
Acronym: Latin-MH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Universidad Peruana Cayetano Heredia (Other); London School of Hygiene and Tropical Medicine (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Paulo Rossi Menezes, Full Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1U19MH098780-01 SP; 1U19MH098780-01 (NIH)
Record Dates: First submitted 2016-03-31; First posted 2016-07-27 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Depression; Diabetes; Hypertension
Keywords: depression; mobile technology; community trial
MeSH Terms: conditions — Depression; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONEMO (Experimental): Participants will be offered a behavioral activation-based intervention delivered by an applicative for smartphones (CONEMO), which encourages them to be more active and to incorporate more activities in their everyday life.
  Primary care nurses will train participants to use the CONEMO app, monitor patients' adherence to CONEMO, calling patients when they are non-adherent, and give technical support when necessary. They will be supervised by clinical psychologists.
  Primary care teams are informed of participants' depression level and deliver usual care according to clinical protocols, including the assessment for the need of antidepressant medication.
  Interventions: Behavioral: CONEMO
- ENHANCED USUAL CARE (No Intervention): The primary care teams are informed of the participants' depression level and can deliver usual care according to clinical protocols, including the assessment for the need of antidepressant medication. This is considered enhanced usual care because the teams are notified about participants' level of depressive symptomatology, which otherwise might go undetected, and then decide about the best way to handle with patients' needs related to their depressive symptomatology.

INTERVENTIONS:
Behavioral: CONEMO — The study intervention has two components: the smartphone application CONEMO and primary care nurses monitoring patients' adherence to the intervention. CONEMO is a 6-week low-intensity behavior activation program delivered in 18 sessions that include messages related to the treatment goals, motivating them to do certain activities, helping to select and plan activities and messages related to psychological skills that facilitate the incorporation of activities in everyday life and to tackle obstacles that hinder patients to be more active. Primary care nurses are responsible for training participants to use the CONEMO app, monitoring patients' adherence to CONEMO, calling patients when they are non-adherent, and giving technical support when necessary.
  Arms: CONEMO

SUMMARY:
Background: Depression is a usual comorbid event associated to chronic diseases, such as hypertension and diabetes, constituting an important public health problem, with negative consequences for patients' quality of life and self-care, as well as for compliance with medical treatment. In low and middle income countries depression is often unrecognized and untreated, and there is a lack of human resources to treat depression and other mental problems in these health care systems.

Aim: The present study aims to test a 6 week low-intensity psychological intervention (CONEMO) delivered via an applicative for smartphones for people with depressive symptoms and co-morbid diabetes and/or hypertension recruited in primary health care units, in São Paulo (Brazil).

DETAILED DESCRIPTION:
Epidemiologic research has clearly established the significant public health importance of mental disorders in low- and middle-income countries (LMIC) and their chronic nature. Among mental disorders, depression has become a major problem as a single condition and, more often, as part of complex clinical pictures in which multiple conditions and risk factors are combined.

There is substantial co-morbidity between depression and chronic physical conditions, and outcome of both conditions is impaired when there is this co-morbidity. Most of the disease burden in LA is now explained by chronic diseases, including depression, cardio-vascular diseases -mostly hypertension related- and diabetes. Despite the public health impact of depression, it often goes unrecognized and untreated. One factor for this treatment gap is the lack of financial and human resources. The limited mental health resources available in LMIC are often not optimally distributed either. Funds and trained personnel are typically allocated in tertiary health care services, such as psychiatric hospitals.

Therefore, any short- and medium-term efforts to develop, evaluate, and disseminate effective mental health interventions in LMIC must adapt to these severe workforce, resource limitations, and inequities. The mental health field needs to consider developing self-help automated interventions that can reach people where there are no health care providers. This can be partially addressed through two strategies: 1) increasing effective self-management; and 2) through task-shifting roles to less specialized but appropriately trained health workers.

We are conducting a community cluster randomized trial with individuals with chronic diseases (hypertension and/or diabetes) and symptoms of depression, attending primary care clinics in São Paulo, Brazil. Participating clinics (20) will be randomly allocated to have their nurse assistants trainned and supervised to monitor an intervention based on behavior activation (experimental group) delivered by an applicative for smartphones (CONEMO) or to receive routine care (control group). The focus of this project is on patients helping themselves through the use of resources that provide continuous advice, support, and motivation. However, studies suggest that depressed patients left alone with their own devices fail to make good use of self-help interventions. Nurse assistants will assist participants by a web-based automated interface connected to the smartphone application (CONEMO) and will receive supervision in this task once a week.

Method:

CONEMO is a cluster randomized controlled trial conducted with 880 chronic patients who present diabetes and/ or hypertension and with depression, receiving health care in 20 Primary Care Units with Family Health Program in Sao Paulo, Brazil. Of these, half (10) will deliver the intervention CONEMO and half (10) will deliver usual care.

The intervention, based in behavior activation, is delivered by a smartphone and monitored by health professionals (nurse assistants) working at the primary care unit responsible for the care of the patient. The CONEMO intervention is based on behavior activation and is delivered by an applicative for smartphones 3 times a week during 6 weeks, with a total of 18 sessions. A nurse assistant mediates this intervention, motivating the patient and monitoring his/her performance. Intensity of depressive symptoms and suicidal ideation is assessed by research assistants using the PHQ-9 and standardized protocols for suicidal risk at baseline, 3- and 6-month follow-ups.

The primary outcome is remission of depressive symptoms 3 months after inclusion in the study. Secondary outcomes include remission of depressive symptoms at 6 months after inclusion, social support, quality of life, compliance to medication, suicidal ideation and activities performed.

The effectiveness and cost-effectiveness of the intervention will be assessed with intention-to-treat analysis, using the clinical outcome and the assessment of quality of life (EQ-5D) 3 and 6 months after inclusion in the trial and the use of health services.

Primary Outcome Measures:

Patient Health Questionnaire (PHQ-9) score 3 months after inclusion in the study.

A 50% reduction in the PHQ-9 score from baseline will be considered success.

Secondary Outcome Measures:

Depression - Patient Health Questionnaire (PHQ-9), Quality of life-EQD5, Adherence to medication-Morisky; Social functioning- WHODAS, Daily activities (BADS).

Time Frame: 6 months after inclusion in the study. A 50% reduction on the PHQ-9 score from baseline will be considered success.

Cost effectiveness measures (3 and 6 months). Use of health services and medication. General Quality of life (EQ-5D).

Process evaluation:

Data collected in the interviews with participants and Nurse Assistants about CONEMO system.

ELIGIBILITY:
Inclusion Criteria:

* Attending one of 20 selected primary care clinics
* Clinical diagnosis of diabetes and/or hypertension
* Presenting with depressive symptoms (PHQ-9 ≥10)

Exclusion Criteria:

* Moderate to high suicidal risk (assessed with a standardized protocol)
* Not able to read

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with 50% reduction in PHQ-9 score a 3-month assessment | 3 months after enrollment
  Presence and severity of depressive symptoms is measured with the PHQ-9. A 50% reduction in PHQ-9 score at 3-month assessment as compared to PHQ-9 score at baseline will be considered as treatment success.

SECONDARY OUTCOMES:
Number of participants with 50% reduction in PHQ-9 score a 6-month assessment | 6 months after enrollment
  Presence and severity of depressive symptoms is measured with the PHQ-9. A 50% reduction in PHQ-9 score at 6-month assessment as compared to PHQ-9 score at baseline will be considered as treatment success.
Improvement in scores for Quality of Life, as measured by the EQD5 | 3 and 6 months after enrollment
  Quality of life is measured with the EQ-5D, a standardized instrument that investigates 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Proportion of participants who improve adherence to diabetes or hypertension medications, evaluated by the Morisky questionnaire | 3 and 6 months after enrollment
  proportion of patients who improve adherence to diabetes or hypertension medication 3 and 6 months after enrollment, as compared to baseline, using the Morisky Medication Adherence Scale (MMAS-4). The distribution of MMAS-4 scores according to the level of medication adherence is: High adherence (0), Medium adherence (1-2) and Low adherence.
Number of medical consultations, hospitalizations, and visits to the primary care team | 3 and 6 months after enrollment
  Data on the use of health services will be collected at baseline, 3-month and six-month follow-up. At each assessment, information about medical consultations, hospitalizations, and visits to the primary care team will be obtained with a standardized questionnaire.
Proportion of participants who improve level of activity, as evaluated by the short form of the Behavioral Activation for Depression Scale (BADS) | 3 and 6 months after enrollment
  Level of daily activity: assessed at baseline, 3-month, and 6-month follow-up visits using the short form of the Behavioral Activation for Depression Scale BADS. It is a 9-item scale used to measure the frequency of activation and avoidance behaviors hypothetically underlying depression mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Araya, PhD, Principal Investigator — London School of Medicine; Lisa Colpe, PhD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
One year after the end of the trial data will be available under request

REFERENCES:
- [Derived] Claro HG, Menezes PR, Fernandes IF, Seward N, Miranda JJ, Saidel MGB, Baquete AGL, Daley KL, Aschar S, Cruz DV, Castro HCM, Rocha T, Quayle J, Peters TJ, Araya R. Do baseline participant characteristics impact the effectiveness of a mobile health intervention for depressive symptoms? A post-hoc subgroup analysis of the CONEMO trials. Braz J Psychiatry. 2024;46:e20233172. doi: 10.47626/1516-4446-2023-3172. Epub 2024 Jan 30. PMID 38345934
- [Derived] Vera Cruz Dos Santos D, Coelho de Soarez P, Cavero V, U Rocha TI, Aschar S, Daley KL, Garcia Claro H, Abud Scotton G, Fernandes I, Diez-Canseco F, Brandt LR, Toyama M, Martins Castro HC, Miranda JJ, Araya R, Quayle J, Rossi Menezes P. A Mobile Health Intervention for Patients With Depressive Symptoms: Protocol for an Economic Evaluation Alongside Two Randomized Trials in Brazil and Peru. JMIR Res Protoc. 2021 Oct 13;10(10):e26164. doi: 10.2196/26164. PMID 34643538
- [Derived] Araya R, Menezes PR, Claro HG, Brandt LR, Daley KL, Quayle J, Diez-Canseco F, Peters TJ, Vera Cruz D, Toyama M, Aschar S, Hidalgo-Padilla L, Martins H, Cavero V, Rocha T, Scotton G, de Almeida Lopes IF, Begale M, Mohr DC, Miranda JJ. Effect of a Digital Intervention on Depressive Symptoms in Patients With Comorbid Hypertension or Diabetes in Brazil and Peru: Two Randomized Clinical Trials. JAMA. 2021 May 11;325(18):1852-1862. doi: 10.1001/jama.2021.4348. PMID 33974019
- [Derived] Rocha TIU, Aschar SCAL, Hidalgo-Padilla L, Daley K, Claro HG, Martins Castro HC, Dos Santos DVC, Miranda JJ, Araya R, Menezes PR. Recruitment, training and supervision of nurses and nurse assistants for a task-shifting depression intervention in two RCTs in Brazil and Peru. Hum Resour Health. 2021 Feb 5;19(1):16. doi: 10.1186/s12960-021-00556-5. PMID 33546709